CLINICAL TRIAL: NCT01524055
Title: CO2 Insufflation During Single-Balloon-Enteroscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Albert Schweitzer Hospital (Other); Nuovo Ospedale Civile S.Agostino Estense (Other); Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18052011; CO2 Insufflation During SBE (Other: University Hospital of Muenster)
Record Dates: First submitted 2011-12-14; First posted 2012-02-01 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Single-Balloon Enteroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Air (Other): Air as insufflation gas during single-balloon enteroscopy.
  Interventions: Device: Single-Balloon-Enteroscopy with Air as insufflation gas.
- CO2 (Other): CO2 as insufflation gas during single-balloon enteroscopy.
  Interventions: Device: Single-Balloon-Enteroscopy with CO2 as insufflation gas.

INTERVENTIONS:
Device: Single-Balloon-Enteroscopy with Air as insufflation gas. — Single-Balloon-Enteroscopy will be performed using Air as insufflation gas to inflate the intestine for complete examination.
  Other Names: SIF-Q180, Olympus Optical, Tokyo, Japan
  Arms: Air
Device: Single-Balloon-Enteroscopy with CO2 as insufflation gas. — Single-Balloon-Enteroscopy will be performed using CO2 as insufflation gas to inflate the intestine for complete examination.
  Other Names: SIF-Q180, Olympus Optical, Tokyo, Japan
  Arms: CO2

SUMMARY:
Double-balloon enteroscopy (DBE) was introduced 2001 for visualizing the entire small bowel. In 2008, a novel balloon-assisted enteroscope system has been developed using only a single balloon (single-balloon enteroscope, SBE). SBE was designed to facilitate diagnosis and treatment of the small bowel. The investigators could demonstrate the both endoscopic procedures are equally suitable in the clinical routine. In both balloon-assisted endoscopic procedures (balloon-assisted enteroscopy (BAE)) it is mandatory to insufflate gas into the bowel to secure good visualization. All endoscopes used for GI endoscopy provide a gas insufflation unit. Currently, many endoscopy units use air for this purpose. The use of air, however, is far from ideal for insufflation in GI endoscopy. During and after GI endoscopy, significant amounts of air are usually retained in the bowel segment inspected. This air has to pass the GI tract and exit physiologically through the rectum. Thus, abdominal pain and discomfort during and after the examination due to the retention of air have been shown to be very common during and after endoscopic procedures. Carbon dioxide gas (CO2), unlike air, is rapidly absorbed from the bowel. Within minutes, several liters of CO2 can be absorbed from the GI tract. The use of CO2 has been shown to result in more comfortable examinations in both colonoscopy and flexible sigmoidoscopy in several randomized trials. In these studies, CO2 insufflation had almost completely reduced procedure-related pain and discomfort.

In 2007, the investigators could demonstrate the advantages of CO2-Insufflation in DBE. Another group confirmed our findings. To our knowledge, no study has been performed investigating the use of CO2 in SBE.

The aim of the present study is to examine whether CO2 insufflation leads to a reduction of abdominal pain in SBE patients. Furthermore, the investigators want to investigate if CO2 insufflation facilities a deeper intubation of the endoscope, as shown for the DBE technique.

DETAILED DESCRIPTION:
Double-balloon enteroscopy (DBE) was introduced 2001 for visualizing the entire small bowel. 2008, a novel balloon enteroscope system has been developed using only a single balloon (single-balloon enteroscope, SBE). SBE was designed to facilitate diagnosis and treatment of the small bowel. We could demonstrate the both endoscopic procedures are equally suitable in the clinical routine. In both balloon-assisted endoscopic procedures (balloon-assisted enteroscopy (BAE)) it is mandatory to insufflate gas into the bowel to secure good visualization. All endoscopes used for GI endoscopy provide a gas insufflation unit. Currently, many endoscopy units use air for this purpose. The use of air, however, is far from ideal for insufflation in GI endoscopy. During and after GI endoscopy, significant amounts of air are usually retained in the bowel segment inspected. This air has to pass the GI tract and exit physiologically through the rectum. Thus, abdominal pain and discomfort during and after the examination due to the retention of air has been shown to be very common during and after endoscopic procedures. Carbon dioxide gas (CO2), unlike air, is rapidly absorbed from the bowel. Within minutes, several liters of CO2 can be absorbed from the GI tract. The use of CO2 has been shown to result in more comfortable examinations in both colonoscopy and flexible sigmoidoscopy in several randomized trials. In these studies, CO2 insufflation almost completely reduced procedure-related pain and discomfort.

In 2007, we could demonstrate the advantages of CO2-Insufflation in DBE. Another group confirmed our findings. To our knowledge, no research has been performed investigating the use of CO2 in SBE.

BAE is a long-lasting procedure. Large volumes of air are insufflated during the procedure, leading to significant distension of the small bowel during and after the examination.

One of the main technical difficulties in BAE is the formation of small bowel loops and sharp angels during deep intubation of the endoscope. These loops and angels are the major restriction to deep intubation of the endoscope. Loops and sharp angels are more pronounced in air-distended bowel segments.

The aim of the present study is to examine whether CO2 insufflation leads to a reduction of abdominal pain in SBE patients. Furthermore, we want to investigate if CO2 insufflation facilities a deeper intubation of the endoscope, as shown for the DBE technique.

Hypothesis

1. The use of CO2 in SBE leads to a reduction in abdominal pain for the patient when compared with the use of air.
2. The use of CO2 in SBE leads to deeper intubation when compared to air insufflation.

The study is designed as a two-center randomized controlled trial. Randomization to the two groups (CO2 vs. air insufflation) is performed of individual participant basis.

Randomization to the two groups (CO2 vs air insufflation) is performed on basis of the individual participant. Equally large groups are randomized, using block randomization (blocks of six patients) for each of the participating centers. Randomization (using SPSS statistical software package) is performed by an independent researcher, who is not part of the SBE team.

Individuals eligible for inclusion are patients referred for SBE at the trial centers who do not fulfill one of the following exclusion criteria:

* Age under 16 years
* Inability to understand information for participation
* Refusal of participation

All eligible individuals are informed about the nature of the study. All individuals provide written informed consent before entering the trial. Patients who do not wish to participate in the present trial are treated according to standard procedures (using air insufflation).

All procedures are performed by experienced endoscopists. Both patients and endoscopists are blinded with regard to type of gas used for any particular patient.

Sedation is performed according to current standards at the centers. Single-balloon procedure SBE is performed using the SBE endoscope system (SIF-Q180, Olympus Optical, Tokyo, Japan), as described in the literature 2-4.

Gas insufflation CO2 is insufflated using EZEM equipment (or other, to be specified). Air is insufflated using the ordinary air inlet system of the endoscope rack. The air inlet button is hidden from the view of the endoscopist to prevent unblinding (technical details to be specified in cooperation with company).

For evaluation of pain and discomfort, a questionnaire is used to classify patient pain during and after the procedure. Visual analogue scales (100-mm) are used to quantify abdominal pain during the examination and at 1, 3, 6, and 24 hours after the procedure, as validated in recent studies7,8. The questionnaire is given to every participant after the procedure, to be filled in the next day.

All procedure parameters of interest (e.g. duration, depth of insertion, use of sedatives) are registered by the endoscopist immediately after the examination using the existing GI lab databases.

Ethics The regional ethics committees of the participating centers will be asked for approval of the study protocol.

Power analysis: a 25% improvement of intubation depth is considered to be clinically important to detect. On the basis of our DBE-CO2-study9, power calculation was conducted determining the size of the study (n=66).

Ownership data are owned by the respective centers. Publication of the study results is planned in a peer-reviewed journal. Philipp Lenz and Dirk Domagk will co-ordinate study design, data generation and analysis and a first manuscript draft.

Budget: All procedures in the present study are performed in ordinary patients, with ordinary staff and endoscopists. Therefore, no extra costs occur for personal.

ELIGIBILITY:
Inclusion Criteria:

• Indication for Single-Balloon-Enteroscopy

Exclusion Criteria:

* Age under 16 years
* Inability to understand information for participation
* Refusal of participation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Intubation depth | 2h
  The endoscopists estimate the depth of intubation during each examination using a recently described and validated technique.

SECONDARY OUTCOMES:
Number of participants with severe adverse events related to the endoscopic procedure | 48h
  SAE related to the endoscopic procedure: number of participants with severe adverse events as a measure of safety and tolerability.
Abdominal pain on on the visual analog scale | 24h
  For evaluation of pain and discomfort, a questionnaire (Pain scores on the visual analog scale) is used to classify patient pain during and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Domagk, M.D., PhD, Principal Investigator — Department of Medicine B
Locations (4):
- Germany (2):
  - University Hopstial of Muenster, Department of Medicine B, Münster
  - HELIOS Albert-Schweitzer-Hospital, Northeim
- Italy (2):
  - Gastroenterology and Digestive Endoscopy Unit, Nuovo Ospedale Civile S.Agostino-Estense, Baggiovara Di Modena
  - San Giovanni Battista University Teaching Hospital, Department of Medicine, Division of Gastroenterology 2, Torino

REFERENCES:
- [Background] Yamamoto H, Sekine Y, Sato Y, Higashizawa T, Miyata T, Iino S, Ido K, Sugano K. Total enteroscopy with a nonsurgical steerable double-balloon method. Gastrointest Endosc. 2001 Feb;53(2):216-20. doi: 10.1067/mge.2001.112181. PMID 11174299
- [Background] Hartmann D, Eickhoff A, Tamm R, Riemann JF. Balloon-assisted enteroscopy using a single-balloon technique. Endoscopy. 2007 Feb;39 Suppl 1:E276. doi: 10.1055/s-2007-966616. Epub 2007 Oct 24. No abstract available. PMID 17957636
- [Background] Tsujikawa T, Saitoh Y, Andoh A, Imaeda H, Hata K, Minematsu H, Senoh K, Hayafuji K, Ogawa A, Nakahara T, Sasaki M, Fujiyama Y. Novel single-balloon enteroscopy for diagnosis and treatment of the small intestine: preliminary experiences. Endoscopy. 2008 Jan;40(1):11-5. doi: 10.1055/s-2007-966976. Epub 2007 Dec 4. PMID 18058613
- [Background] Domagk D, Mensink P, Aktas H, Lenz P, Meister T, Luegering A, Ullerich H, Aabakken L, Heinecke A, Domschke W, Kuipers E, Bretthauer M. Single- vs. double-balloon enteroscopy in small-bowel diagnostics: a randomized multicenter trial. Endoscopy. 2011 Jun;43(6):472-6. doi: 10.1055/s-0030-1256247. Epub 2011 Mar 7. PMID 21384320
- [Background] Hussein AM, Bartram CI, Williams CB. Carbon dioxide insufflation for more comfortable colonoscopy. Gastrointest Endosc. 1984 Apr;30(2):68-70. doi: 10.1016/s0016-5107(84)72319-4. PMID 6425108
- [Background] Bretthauer M, Thiis-Evensen E, Huppertz-Hauss G, Gisselsson L, Grotmol T, Skovlund E, Hoff G. NORCCAP (Norwegian colorectal cancer prevention): a randomised trial to assess the safety and efficacy of carbon dioxide versus air insufflation in colonoscopy. Gut. 2002 May;50(5):604-7. doi: 10.1136/gut.50.5.604. PMID 11950803
- [Background] Stevenson GW, Wilson JA, Wilkinson J, Norman G, Goodacre RL. Pain following colonoscopy: elimination with carbon dioxide. Gastrointest Endosc. 1992 Sep-Oct;38(5):564-7. doi: 10.1016/s0016-5107(92)70517-3. PMID 1397911
- [Background] Sumanac K, Zealley I, Fox BM, Rawlinson J, Salena B, Marshall JK, Stevenson GW, Hunt RH. Minimizing postcolonoscopy abdominal pain by using CO(2) insufflation: a prospective, randomized, double blind, controlled trial evaluating a new commercially available CO(2) delivery system. Gastrointest Endosc. 2002 Aug;56(2):190-4. doi: 10.1016/s0016-5107(02)70176-4. PMID 12145595
- [Background] Domagk D, Bretthauer M, Lenz P, Aabakken L, Ullerich H, Maaser C, Domschke W, Kucharzik T. Carbon dioxide insufflation improves intubation depth in double-balloon enteroscopy: a randomized, controlled, double-blind trial. Endoscopy. 2007 Dec;39(12):1064-7. doi: 10.1055/s-2007-966990. PMID 18072057
- [Background] Hirai F, Beppu T, Nishimura T, Takatsu N, Ashizuka S, Seki T, Hisabe T, Nagahama T, Yao K, Matsui T, Beppu T, Nakashima R, Inada N, Tajiri E, Mitsuru H, Shigematsu H. Carbon dioxide insufflation compared with air insufflation in double-balloon enteroscopy: a prospective, randomized, double-blind trial. Gastrointest Endosc. 2011 Apr;73(4):743-9. doi: 10.1016/j.gie.2010.10.003. Epub 2011 Jan 14. PMID 21237455
- [Derived] Lenz P, Meister T, Manno M, Pennazio M, Conigliaro R, Lebkucher S, Ullerich H, Schmedt A, Floer M, Beyna T, Lenze F, Domagk D. CO2 insufflation during single-balloon enteroscopy: a multicenter randomized controlled trial. Endoscopy. 2014 Jan;46(1):53-8. doi: 10.1055/s-0033-1359041. Epub 2013 Dec 18. PMID 24353124